CLINICAL TRIAL: NCT05147831
Title: Effectiveness of Remote Ischemic Preconditioning for Prevention of Contrast Induced Acute Kidney Injury in Patients Undergoing Coronary Angiograms.
Acronym: RIP-CI-AKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21-0280
Record Dates: First submitted 2021-11-26; First posted 2021-12-07 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Contrast-induced Acute Kidney Injury (CI-AKI) Following Coronary Angiogram (CI-AKI); Contrast-induced Nephropathy Following Coronary Angiogram (CIN)
Keywords: Contrast-induced acute kidney injury (CI-AKI); Coronary angiogram; Contrast-induced nephropathy (CIN)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning Protocol (Experimental)
  Interventions: Other: Remote Ischemic Preconditioning
- Sham Preconditioning Protocol (No Intervention)

INTERVENTIONS:
Other: Remote Ischemic Preconditioning — Place blood pressure cuff around upper, non-dominant arm (e.g. upper left arm in a right-handed patient). Inflate blood pressure cuff to a pressure set at 50 mmHg higher than baseline systolic BP to induce ischemia of arm for 5 minutes. Completely deflate blood pressure cuff to allow for 5 minutes of reperfusion. Subjects would undergo 4 cycles of ischemia and reperfusion,
  Arms: Remote Ischemic Preconditioning Protocol

SUMMARY:
The use of imaging is increasing in clinical practice, either for diagnosis or intervention. In these imaging processes, contrast medium (CM) is widely used. However, CM administration can induce contrast-induced nephropathy (CI-AKI). CI-AKI is the third most common cause of renal insufficiency, and its incidence varies from 2% to 50% depending on patient risk factors; in addition, studies have shown that CI-AKI occurs in 2% to 25% of patients undergoing coronary intervention. CI-AKI is associated with significant mortality and morbidity in patients undergoing coronary angiography or other diagnostic contrast studies. We assessed the latest promising evidence on the ability of remote ischemic preconditioning (RIPC) to reduce the incidence of CI-AKI in patients undergoing Coronary Angiogram (CA) or diagnostic contrast studies such as CT angiogram, while at the same time being a non-invasive, low cost, easy, and safe method with absence of adverse effects. However, more randomized controlled trials are needed to confirm these preliminary results.

The aim of this study is to minimize the incidence of CI-AKI at the University of Texas Medical Branch (UTMB). If found to be an effective method, RIPC would help minimize the incidence of CI-AKI in all institutions across the globe, who would adopt this intervention.

The primary objective: i) reduce the rise in creatinine to < 0.5 mg/dL post-CA in moderate to high risk patients and ii) reduce the incidence of renal replacement therapy post-CA in moderate to high risk patients; iii) we also aim to establish that RIPC is safe and effective.

We hypothesize that the use of RIPC, when added to standard medical therapy (pre-and post-CA hydration), will mitigate the effects of contrast on the renal vasculature and lessen the incidence of CI-AKI in moderate to high risk patients at the University of Texas Medical Branch.

The use of iodinated contrast to visually enhance target vasculature is a widely used diagnostic technique that is performed daily at UTMB, and around the world, for the diagnosis and management of a variety of conditions. A common complication of this procedure is acute kidney injury (AKI), generally referred to as contrast-induced nephropathy (CI-AKI). This complication can range from an isolated rise in serum creatinine to severe renal dysfunction necessitating renal replacement therapy. The incidence of CI-AKI has been reported as approximately 2-50%, depending upon the definition and sensitivity of assay employed to assess GFR in the hospital setting. In addition, CI-AKI is associated with significant mortality and morbidity. If proven to be beneficial, RIPC will bring about a reduction in incidence of CI-AKI, and thus help to reduce hospitalization and mortality from renal etiology following a given contrast procedure.

DETAILED DESCRIPTION:
The use of imaging is increasing in clinical practice, either for diagnosis or intervention. In these imaging processes, contrast medium (CM) is widely used. However, CM administration can induce contrast-induced nephropathy (CI-AKI). CI-AKI is the third most common cause of renal insufficiency, and its incidence varies from 2% to 50% depending on patient risk factors; in addition, studies have shown that CI-AKI occurs in 2% to 25% of patients undergoing coronary intervention. CI-AKI is associated with significant mortality and morbidity in patients undergoing coronary angiography or other diagnostic contrast studies. We assessed the latest promising evidence on the ability of remote ischemic preconditioning (RIPC) to reduce the incidence of CI-AKI in patients undergoing Coronary Angiogram (CA) or diagnostic contrast studies such as CT angiogram, while at the same time being a non-invasive, low cost, easy, and safe method with absence of adverse effects. However, more randomized controlled trials are needed to confirm these preliminary results.

The aim of this study is to minimize the incidence of CI-AKI at the University of Texas Medical Branch (UTMB). If found to be an effective method, RIPC would help minimize the incidence of CI-AKI in all institutions across the globe, who would adopt this intervention.

The primary objective: i) reduce the rise in creatinine to < 0.5 mg/dL post-CA in moderate to high risk patients and ii) reduce the incidence of renal replacement therapy post-CA in moderate to high risk patients; iii) we also aim to establish that RIPC is safe and effective.

We hypothesize that the use of RIPC, when added to standard medical therapy (pre-and post-CA hydration), will mitigate the effects of contrast on the renal vasculature and lessen the incidence of CI-AKI in moderate to high risk patients at the University of Texas Medical Branch.

The use of iodinated contrast to visually enhance target vasculature is a widely used diagnostic technique that is performed daily at UTMB, and around the world, for the diagnosis and management of a variety of conditions. A common complication of this procedure is acute kidney injury (AKI), generally referred to as contrast-induced nephropathy (CI-AKI). This complication can range from an isolated rise in serum creatinine to severe renal dysfunction necessitating renal replacement therapy. The incidence of CI-AKI has been reported as approximately 2-50%, depending upon the definition and sensitivity of assay employed to assess GFR in the hospital setting. In addition, CI-AKI is associated with significant mortality and morbidity. If proven to be beneficial, RIPC will bring about a reduction in incidence of CI-AKI, and thus help to reduce hospitalization and mortality from renal etiology following a given contrast procedure.

Risk factors for CI-AKI include age > 75, hypotension, CHF, anemia, diabetes, patients with a baseline serum creatinine greater than 1.5 mg /dL and the volume of contrast media used. The presence of underlying renal dysfunction appears to provide particular susceptibility. Although most studies exclude patients with severe renal dysfunction, Rihal et al. report that in patients with a creatinine >3.0 (and GFR < 30) the incidence of CI-AKI was 31%.

Unfortunately, robust strategies to prevent CI-AKI are minimal. Research has examined the use of sodium bicarbonate, adding N-acetylcysteine or holding RAAS (Renin-angiotensin-aldosterone system) blockers but found all these three strategies ineffective. At this time the only validated strategy to prevent CI-AKI is the use of fluid administration to ensure adequate renal perfusion. Pre- and post-procedure intravenous fluid administration is currently considered standard of care. In one study involving 408 patients with intact renal function receiving isotonic saline (NS) (1cc/kg/h before percutaneous angiography and 24 hours after) the incidence of CI-AKI within the following 3 days was 21% in the group without NS and 11% in the NS+ group (p=0.016). Further, CI-AKI was associated with increased risk of death (15.2% vs 2.8%; p<0.0001) and need for renal replacement therapy (13.4% vs 0%; p<0.0001). In another trial involving 216 patients, pre- and post-procedure hydration reduced the incidence of CI-AKI in the hydrated group versus the non-hydrated control group 20.4% versus 35.2%, p< 0.05). These results were confirmed in the POSEIDON trial which also showed that a LVEDP (left ventricular end-diastolic pressure) guided hydration strategy for the prevention of CI-AKI results in an even greater relative and absolute risk reduction in contrast nephropathy in comparison to the standard hydration strategy.

The pathophysiology of CI-AKI is thought to involve renal artery vasoconstriction and the development of reactive oxygen species which leads to direct renal oxidative stress and ischemic injury.

Kidney Disease Improving Global Outcome (KDIGO) defines CI-AKI as an increase in serum creatinine level ≥0.5 mg/dl or >25% compared with the baseline value within a period of 48-72 hours after contrast media (CM) administration.

The definition of Remote Ischemic Preconditioning is not as simple. According to a pathophysiologic concept, repeated short duration ischemia in an organ induces a ''resistance'' to a later prolonged ischemia. That is, a brief period of ischemia induces endogenous protective mechanisms that increase tissue tolerance to subsequent lethal ischemia. This is a physiological adaptive mechanism of protection of tissues faced to hypoperfusion, which has therapeutic potential when ischemia-reperfusion is induced in a targeted way. In 1982, this mechanism called ischemic preconditioning (IPC) was highlighted for the first time on canine models in myocardial infarction. In experiments, cycles of alternating ischemia and reperfusion were applied to dogs by using a balloon to occlude a coronary artery. This allowed the prevention of necrotic myocardial territories. These results have opened prospects on a possible use of this method of preconditioning for myocardial protection as well as preconditioning for renal protection in humans.

Our remote ischemic preconditioning protocol would comprise four (4) cycles of 5 min of ischemia followed by 5 min of reperfusion for the experimental group. The BP cuff would be placed around the upper non-dominant arm (e.g upper left arm in a right-handed patient) and inflated to a pressure set at 50 mmHg higher than baseline systolic BP to induce transient ischemia followed by subsequent deflation to ensure 5 minutes of reperfusion in the RIPC group. The absence of distal pulse would be confirmed with Doppler evaluation or palpation of the radial and ulnar artery.

In the control group, sham preconditioning would be performed by inflating an upper-arm blood pressure cuff to diastolic pressure levels and then deflating the cuff to 10 mm Hg below diastolic pressure for 5 minutes to maintain nonischemic upper-arm compression for blinding purposes with regard to the patients; this will be followed by complete deflation of cuff for 5 minutes. Again a total of four cycles would be ensured. In individuals presenting with BMI > 30 kg/m2 , a dedicated blood pressure cuff for obese patients will be used. Time from RIPC to the procedure (either CA or diagnostic contrast study) will be within <120 min in all studies.

The patients will be randomly assigned in a 1:1 ratio to either the control group or RIPC group. Randomization will be performed by data analysis software, which would determine whether the patient would fall under the RIPC arm vs Sham-procedure arm.

All patients will receive standard care for patients with impaired renal function undergoing CA:

Recommended hydration will consist of saline 0.9% solution infusion at a rate of 1 mL/Kg/h for 12 hours prior to contrast medium injection and up to 12 hours thereafter, unless there is evidence of fluid overload thus contraindicating further fluid administration. Metformin, angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, diuretics, and non-steroidal anti-inflammatory drugs will be discontinued at least 24 hours before the angiography. Blood samples for basic metabolic panel (BMP) would be drawn prior to coronary intervention/diagnostic contrast study and repeated 48-72 hrs following contrast medium administration. A final BMP would be checked at 6 weeks after contrast procedure.

Following IRB approval, studies will begin with a target of including 300 patients in the study, with a tentative timeline of three (3) years. We will obtain BMPs on the day of the procedure (to document baseline creatinine), and then repeat 48-72 hrs after CA/diagnostic contrast studies. No additional visits would be required apart from a visit to the phlebotomist for getting the BMP checked within 48-72 hrs and another visit for repeat BMP check at 6 weeks. Almost all of our patients who undergo CA will have a follow-up appointment with their PCP in the next 3-7 days, but no extra visits are required for the study purpose. No extra costs on the part of the patient would be necessary.

Our intervention group- remote ischemic preconditioning group- would be subject to four (4) cycles of 5 min of ischemia followed by 5 min of reperfusion for the experimental group. The BP cuff would be placed around the upper non-dominant arm (e.g upper left arm in a right-handed patient) and inflated to a pressure set at 50 mmHg higher than baseline systolic BP to induce transient ischemia followed by subsequent deflation to ensure 5 minutes of reperfusion in the RIPC group. The absence of distal pulse would be confirmed with Doppler evaluation or palpation of the radial and ulnar artery.

In the control group, sham preconditioning would be performed by inflating an upper-arm blood pressure cuff to diastolic pressure levels and then deflating the cuff to 10 mm Hg below diastolic pressure for 5 minutes to maintain nonischemic upper-arm compression for blinding purposes with regard to the patients; this will be followed by complete deflation of cuff for 5 minutes. Again a total of four cycles would be ensured. In individuals presenting with BMI > 30 kg/m2 , a dedicated blood pressure cuff for obese patients will be used. Time from RIPC to the procedure (either CA or diagnostic contrast study) will be within <120 min in all studies.

In addition to our above mentioned intervention (RIPC), all patients will receive standard of care for patients with impaired renal function undergoing CA as mentioned below (No.1 and No.2) :-

No.1: Recommended hydration will consist of saline 0.9% solution infusion at a rate of 1 mL/Kg/h for 12 hours prior to contrast medium injection and up to 12 hours thereafter, unless there is evidence of fluid overload thus contraindicating further fluid administration.

No.2: Metformin, angiotensin-converting enzyme inhibitors, angiotensin II receptor blockers, diuretics, and non-steroidal anti-inflammatory drugs will be discontinued at least 24hours before the angiography.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients undergoing an interventional or diagnostic radiological procedure in which they receive intravascular contrast, including patients undergoing coronary angiogram +/- percutaneous coronary intervention (PCI) for all clinical indications except those indicated for primary PCI due to STEMI
* (2) patients presenting with a renal clearance in the range of less than 60 ml/min/1.73 m2 but not declared ESRD
* (3) Patients who are not yet recruited for other pharmacological or medical device clinical trials.

Exclusion Criteria:

* (1) Age <18 years
* (2) Patient on hemodialysis or peritoneal dialysis
* (3) Simultaneous participation in another interventional study
* (4) Percutaneous coiling/embolization procedures of the kidney
* (5) Impossibility to perform RIPC, caused by pathology in both arms (e.g. dystrophy, recent trauma, chronic wounds)
* (6) No written informed consent
* (7) Urgent angiography in STEMI
* (8) Cardiogenic shock requiring catecholamine infusion
* (9) Systolic blood pressure <80 mmHg
* (10) Intra-aortic balloon counter-pulsation
* (11) Contrast medium injection within the previous 30 days
* (12) Expected impossibility to obtain follow-up data at 6-week follow-up
* (13) Patients with Raynaud's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Serum Creatinine | Patient's serum creatinine would be measured 48-72 hours after coronary angiogram, and re-measured 6 weeks after coronary angiogram.
  The primary outcome would be the incidence of CI-AKI, which is defined as an increment of serum creatinine ≥ 0.5 mg/dL or a relative increase of ≥ 25% over the baseline value within a period of 48-72 hours after contrast medium administration.

SECONDARY OUTCOMES:
Occurrence of re-hospitalization | Within 6 weeks of coronary angiogram
The need for a session of hemodialysis | Within 6 weeks of coronary angiogram
Mortality within 6 weeks of contrast administration | Within 6 weeks of coronary angiogram
Major adverse events at 6 weeks, which would comprise death from all causes, including cardiovascular death, non-fatal infarction, hemofiltration or hemodialysis, and congestive heart failure leading to hospital admission. | Within 6 weeks of coronary angiogram

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas- Medical Branch (UTMB), Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Er F, Nia AM, Dopp H, Hellmich M, Dahlem KM, Caglayan E, Kubacki T, Benzing T, Erdmann E, Burst V, Gassanov N. Ischemic preconditioning for prevention of contrast medium-induced nephropathy: randomized pilot RenPro Trial (Renal Protection Trial). Circulation. 2012 Jul 17;126(3):296-303. doi: 10.1161/CIRCULATIONAHA.112.096370. Epub 2012 Jun 26. PMID 22735306
- [Background] Solomon RJ, Mehran R, Natarajan MK, Doucet S, Katholi RE, Staniloae CS, Sharma SK, Labinaz M, Gelormini JL, Barrett BJ. Contrast-induced nephropathy and long-term adverse events: cause and effect? Clin J Am Soc Nephrol. 2009 Jul;4(7):1162-9. doi: 10.2215/CJN.00550109. Epub 2009 Jun 25. PMID 19556381
- [Background] Rihal CS, Textor SC, Grill DE, Berger PB, Ting HH, Best PJ, Singh M, Bell MR, Barsness GW, Mathew V, Garratt KN, Holmes DR Jr. Incidence and prognostic importance of acute renal failure after percutaneous coronary intervention. Circulation. 2002 May 14;105(19):2259-64. doi: 10.1161/01.cir.0000016043.87291.33. PMID 12010907
- [Background] Chertow GM, Burdick E, Honour M, Bonventre JV, Bates DW. Acute kidney injury, mortality, length of stay, and costs in hospitalized patients. J Am Soc Nephrol. 2005 Nov;16(11):3365-70. doi: 10.1681/ASN.2004090740. Epub 2005 Sep 21. PMID 16177006
- [Background] Lassnigg A, Schmidlin D, Mouhieddine M, Bachmann LM, Druml W, Bauer P, Hiesmayr M. Minimal changes of serum creatinine predict prognosis in patients after cardiothoracic surgery: a prospective cohort study. J Am Soc Nephrol. 2004 Jun;15(6):1597-605. doi: 10.1097/01.asn.0000130340.93930.dd. PMID 15153571
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Piskinpasa S, Altun B, Akoglu H, Yildirim T, Agbaht K, Yilmaz R, Peynircioglu B, Cil B, Aytemir K, Turgan C. An uninvestigated risk factor for contrast-induced nephropathy in chronic kidney disease: proteinuria. Ren Fail. 2013;35(1):62-5. doi: 10.3109/0886022X.2012.741646. Epub 2012 Nov 23. PMID 23176376
- [Background] Rosenstock JL, Bruno R, Kim JK, Lubarsky L, Schaller R, Panagopoulos G, DeVita MV, Michelis MF. The effect of withdrawal of ACE inhibitors or angiotensin receptor blockers prior to coronary angiography on the incidence of contrast-induced nephropathy. Int Urol Nephrol. 2008;40(3):749-55. doi: 10.1007/s11255-008-9368-1. Epub 2008 Apr 26. PMID 18438718
- [Background] Weisbord SD, Gallagher M, Jneid H, Garcia S, Cass A, Thwin SS, Conner TA, Chertow GM, Bhatt DL, Shunk K, Parikh CR, McFalls EO, Brophy M, Ferguson R, Wu H, Androsenko M, Myles J, Kaufman J, Palevsky PM; PRESERVE Trial Group. Outcomes after Angiography with Sodium Bicarbonate and Acetylcysteine. N Engl J Med. 2018 Feb 15;378(7):603-614. doi: 10.1056/NEJMoa1710933. Epub 2017 Nov 12. PMID 29130810
- [Background] Jurado-Roman A, Hernandez-Hernandez F, Garcia-Tejada J, Granda-Nistal C, Molina J, Velazquez M, Albarran A, Tascon J. Role of hydration in contrast-induced nephropathy in patients who underwent primary percutaneous coronary intervention. Am J Cardiol. 2015 May 1;115(9):1174-8. doi: 10.1016/j.amjcard.2015.02.004. Epub 2015 Feb 12. PMID 25759106
- [Background] Luo Y, Wang X, Ye Z, Lai Y, Yao Y, Li J, Liu X. Remedial hydration reduces the incidence of contrast-induced nephropathy and short-term adverse events in patients with ST-segment elevation myocardial infarction: a single-center, randomized trial. Intern Med. 2014;53(20):2265-72. doi: 10.2169/internalmedicine.53.1853. Epub 2014 Oct 15. PMID 25318787
- [Background] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Walsh SR, Boyle JR, Tang TY, Sadat U, Cooper DG, Lapsley M, Norden AG, Varty K, Hayes PD, Gaunt ME. Remote ischemic preconditioning for renal and cardiac protection during endovascular aneurysm repair: a randomized controlled trial. J Endovasc Ther. 2009 Dec;16(6):680-9. doi: 10.1583/09-2817.1. PMID 19995115
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Atanda AC, Olafiranye O. Contrast-induced acute kidney injury in interventional cardiology: Emerging evidence and unifying mechanisms of protection by remote ischemic conditioning. Cardiovasc Revasc Med. 2017 Oct-Nov;18(7):549-553. doi: 10.1016/j.carrev.2017.06.001. Epub 2017 Jun 6. PMID 28610773
- [Background] Savaj S, Savoj J, Jebraili I, Sezavar SH. Remote ischemic preconditioning for prevention of contrast-induced acute kidney injury in diabetic patients. Iran J Kidney Dis. 2014 Nov;8(6):457-60. PMID 25362220
- [Background] Zagidullin NS, Dunayeva AR, Plechev VV, Gilmanov AZ, Zagidullin SZ, Er F, Pavlov VN. Nephroprotective effects of remote ischemic preconditioning in coronary angiography. Clin Hemorheol Microcirc. 2017;65(3):299-307. doi: 10.3233/CH-16184. PMID 27814282
- [Background] Bafna AA, Shah HC. Remote ischemic preconditioning for prevention of contrast-induced nephropathy - A randomized control trial. Indian Heart J. 2020 Jul-Aug;72(4):244-247. doi: 10.1016/j.ihj.2020.04.010. Epub 2020 May 26. PMID 32861377
- [Background] Mayor F, Bilgin-Freiert A, Connolly M, Katsnelson M, Dusick JR, Vespa P, Koch S, Gonzalez NR. Effects of remote ischemic preconditioning on the coagulation profile of patients with aneurysmal subarachnoid hemorrhage: a case-control study. Neurosurgery. 2013 Nov;73(5):808-15; discussion 815. doi: 10.1227/NEU.0000000000000098. PMID 23867300